CLINICAL TRIAL: NCT00081601
Title: An Open-Label Phase 2 Study of Oral CEP-701 in Patients With Asymptomatic Hormone-Refractory Cancer With Rising Prostate Specific Antigen
Brief Title: Study of CEP-701 in Treatment of Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0701a/203/ON/US
Record Dates: First submitted 2004-04-15; First posted 2004-04-19 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate specific antigen; PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — lestaurtinib

INTERVENTIONS:
Drug: CEP-701

SUMMARY:
The purpose of this study is to determine the proportion of patients with a serological prostate specific antigen (PSA) by day 85.

DETAILED DESCRIPTION:
A serological PSA response is defined as a reduction from baseline PSA serum concentration of at least 50%, which is confirmed by a second PSA value 28 or more days later.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 yrs of age
* diagnosis of adenocarcinoma of the prostate
* no detectable metastatic disease as assessed by bone and CT scans
* has increasing serum PSA concentrations
* life expectancy of at least 3 months
* ECOG of 0 or 1
* has been withdrawn from antiandrogen therapy for at least 6 weeks prior to entering screening period

Exclusion Criteria:

* has asymptomatic disease
* has active GI ulceration or bleeding
* has been treated with non-hormonal systemic anticancer therapy or has received radiation within 4 weeks of baseline visit
* bilirubin >2x ULN or ALT or AST >2xULN or serum creatinine >1.5mg/dL
* hemoglobin <9g/dL or platelets below 100,000/uL or ANC below 1500/uL
* receiving treatment for HIV with protease inhibitors
* has had prior malignancy within past 5 yrs with exception of resected basal or squamous cell carcinomas of the skin
* has used investigational drug with previous one month

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-03; Primary Completion 2005-05 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States